CLINICAL TRIAL: NCT00786162
Title: Blood Pressure Self Management for Hypertension & Prehypertension Using an Internet Enabled, Automated Self Management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joseph C. Kvedar, Director, Center for Connected Health, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2006-P-002440
Record Dates: First submitted 2008-10-23; First posted 2008-11-06 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Internet-based hypertension self-management platform
  Interventions: Other: Internet-enabled automated self-management program
- Control (Active Comparator): Installation of BP cuff for communal use at the worksite
  Interventions: Other: BP cuff at workplace

INTERVENTIONS:
Other: Internet-enabled automated self-management program — An internet platform to display blood pressure readings and provide subjects with automated messages and educational information about hypertension management.
  Arms: Intervention
Other: BP cuff at workplace — Provided BP cuff for communal use at the worksite
  Arms: Control

SUMMARY:
The specific aim of the study is to assess the impact of an Internet-enabled, automated, self-management program on blood pressure control of employees of a large local company.

DETAILED DESCRIPTION:
We propose to conduct a randomized controlled trial of an Internet-enabled, automated self-management program. The study will be carried out through six local sites (offices) of a large employer. 3 sites will be intervention sites and 3 will be control sites.

Subjects enrolled from the intervention sites will receive a blood pressure meter and access to an Internet site where they can view their readings, read educational material regarding hypertension management and receive personalized tips and feedback.

Subjects enrolled from the control sites will have access to a blood pressure monitor located at their workplace but will only be provided with basic written information about hypertension at the start of the trial and will receive no feedback.

The trial will run for 6 months from the time of enrollment and the primary outcome measure will be a change in systolic blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Full-time employees of EMC
* Aged 30 to 65 years at time of enrollment
* Any of the following
* A diagnosis of hypertension as defined by one of the following
* Taking an antihypertensive medication
* Being told at least twice by a physician or other health professional that the subject has high blood pressure†
* A BP > 140/90 detected at screening by the research team on 2 separate occasions.
* A diagnosis of prehypertension as defined by a systolic BP between 120-139 or a diastolic BP between 80-89 detected at screening by the research team on 2 separate occasions
* Access to the Internet at work and / or at home

Exclusion Criteria:

* Inability to self-monitor blood pressure due to musculoskeletal or cognitive impairment
* Known secondary cause of hypertension e.g. renal artery stenosis, Cushing's disease.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2007-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure. | 6 months

SECONDARY OUTCOMES:
Assess whether the intervention increases the motivation and self-efficacy of patients managing blood pressure. Assess patient satisfaction with the intervention. Assess the impact of the intervention on healthcare utilization and expenditure | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph C. Kvedar, MD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Watson AJ, Singh K, Myint-U K, Grant RW, Jethwani K, Murachver E, Harris K, Lee TH, Kvedar JC. Evaluating a web-based self-management program for employees with hypertension and prehypertension: a randomized clinical trial. Am Heart J. 2012 Oct;164(4):625-31. doi: 10.1016/j.ahj.2012.06.013. PMID 23067923